CLINICAL TRIAL: NCT03718806
Title: A Phase 1, Open-Label, Study to Investigate Pharmacokinetics, Effect of Food and Safety of a New Immediate-Release Formulation of Zoliflodacin in Healthy Subjects
Brief Title: Study to Investigate Effect of Food and Safety of a New Formulation of Zoliflodacin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STI_ZOLI002
Record Dates: First submitted 2018-10-17; First posted 2018-10-24 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-10

CONDITIONS: Gonorrhea
MeSH Terms: conditions — Gonorrhea | interventions — zoliflodacin

STUDY DESIGN:
Intervention Model Description: It is planned to enroll 2 cohorts of 24 subjects each. Single doses of zoliflodacin (3 g and 4 g) will be assessed within each cohort in a two period cross-over design.
  Cohort 1
  * Regimen A: 3 g zoliflodacin oral suspension; oral administration after an overnight fast
  * Regimen B: 3 g zoliflodacin oral suspension; oral administration with a standardized high calorie, high-fat breakfast
  Cohort 2
  * Regimen C: 4 g zoliflodacin oral suspension; oral administration after an overnight fast
  * Regimen D: 4 g zoliflodacin oral suspension; oral administration with a standardized high calorie, high-fat breakfast
  There will be a minimum washout of 4 days between each period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Regimen A (Experimental): 3 g zoliflodacin oral suspension; oral administration after an overnight fast
  Interventions: Drug: Zoliflodacin
- Regimen B (Experimental): 3 g zoliflodacin oral suspension; oral administration with a standardized high calorie, high-fat breakfast
  Interventions: Drug: Zoliflodacin; Other: high calorie, high fat breakfast
- Regimen C (Experimental): 4 g zoliflodacin oral suspension; oral administration after an overnight fast
  Interventions: Drug: Zoliflodacin
- Regimen D (Experimental): 4 g zoliflodacin oral suspension; oral administration with a standardized high calorie, high-fat breakfast
  Interventions: Drug: Zoliflodacin; Other: high calorie, high fat breakfast

INTERVENTIONS:
Drug: Zoliflodacin — oral suspension; oral administration
Other: high calorie, high fat breakfast — fasted/fed conditions
  Arms: Regimen B; Regimen D

SUMMARY:
This is a phase I, parallel, open-label, randomized, cross-over, single-center study with zoliflodacin administered as granules for oral suspension with or without food.

It is planned to enroll 2 cohorts (Cohorts 1 and 2) of 24 subjects each (48 subjects in total), with the target of achieving data in 20 evaluable subjects per cohort. Single doses of zoliflodacin will be assessed within each cohort in a two period cross-over design.

Each subject will receive one of the following regimens per period, depending on cohort, in a sequence according to the randomization schedule (per cohort, subjects will be randomized immediately before dosing in Period 1), separated by a minimum 4 day washout between each period. The actual length of washout period may change pending emerging PK data.

Cohort 1:

* Regimen A: 3 g zoliflodacin oral suspension; oral administration after an overnight fast
* Regimen B: 3 g zoliflodacin oral suspension; oral administration with a standardized high calorie, high-fat breakfast

Cohort 2

* Regimen C: 4 g zoliflodacin oral suspension; oral administration after an overnight fast
* Regimen D: 4 g zoliflodacin oral suspension; oral administration with a standardized high calorie, high-fat breakfast

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females
2. Age 18 to 55 years of age
3. Body mass index of 18.0 to 30.1 kg/m2
4. Light smokers (less than 5 cigarettes per day) or subjects who are nonsmokers. No smoking (or use of smoking substitute e.g. nicotine patch) is permitted from screening throughout the study
5. Normal arterial BP and HR or, if abnormal, considered not clinically significant by the PI. These will be measured after resting supine for 10 min
6. Registered in agreement with the applicable law on biomedical experimentation
7. Must be willing and able to comply with all study requirements
8. Must be able to understand a written informed consent, which must be obtained prior to initiation of study procedures
9. Must agree to use an adequate method of contraception
10. Must, in the opinion of the investigator, be in good health based upon medical history and physical examination (including vital signs)

Exclusion Criteria:

1. Subjects who have received of zoliflodacin or any IMP in a clinical research study within 5 half-lives or within 30 days prior to first dose. However, in no event, shall the time between last receipt of IMP and first dose be less than 3 months
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
6. Subjects who have regular daily consumption of ≥5 cigarettes daily, or use more than 3 grams (1/8 ounce) of tobacco
7. Excessive intake of caffeine (more than 8 cups daily of beverage containing caffeine)
8. Subjects who have regular daily consumption of more than one liter of xanthine containing beverages
9. Females of childbearing potential who are pregnant or lactating (female subjects must have a negative serum pregnancy test at screening and admission)
10. Have poor venous access that limits phlebotomy
11. Clinically significant abnormal biochemistry, hematology or urinalysis at screening (i.e. aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, creatinine and urea must be within normal ranges) as judged by the investigator at screening and admission (laboratory parameters are listed in Appendix 1)
12. Presence of clinically significant abnormality following review of vital signs, full physical examination and ECG
13. Positive drugs of abuse test result
14. History or presence of any clinically significant acute or chronic disease, including known or suspected human immunodeficiency virus (HIV), HBV or HCV infection
15. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <80 mL/min using the Cockcroft-Gault equation
16. History of cardiovascular, renal, hepatic, chronic respiratory or GI disease, or psychiatric disorder, as judged by the investigator
17. Any clinically important abnormalities in rate, rhythm, conduction or morphology of resting ECG that in the opinion of the PI are clinically significant or may interfere with the interpretation of QTc interval changes
18. Presence of clinical condition or prior therapy which, in the opinion of the Investigator, made the subject unsuitable for the study
19. Subjects who have had surgery (e.g. stomach bypass) or medical condition that might affect absorption of study drug taken orally
20. History of GI ulcer disease, inflammatory bowel disease, indigestion symptoms >3 times a week, or blood in stool in previous 6 months not related to anal trauma
21. Subjects who have had febrile illness within 1 week before the start of the study
22. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
23. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
24. Must not have significant serious skin disease, including rash, food allergy, eczema, psoriasis, or urticaria
25. History of rare hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency
26. History of major surgical procedure or have donated of blood within 12 weeks prior to first dose of study medication or plasma within 7 days prior to first dose of study medication
27. Must not donate blood from clinic admission, throughout the study duration, and for at least 30 days following last dose of study medication
28. Subjects who are taking, or have taken, any prescribed or over-the-counter drug, including antacid drug, (other than 4 g per day acetaminophen, hormone replacement therapy, hormonal contraception) in the 28 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor
29. Use of dietary supplements or herbal remedies (such as St John's Wort), or grapefruit products known to interfere with the CYP3A4 and/or P-gp metabolic pathways during the 14 days before the first dose of trial medication
30. Individuals who have been vaccinated within 4 to 6 weeks before dose administration of the IMP or planned to be vaccinated up to 4 to 6 weeks after dose administration of the IMP
31. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
PK parameter of zoliflodacin : Cmax | Day 3
  the maximum observed concentration of zoliflodacin after a single oral 3 g dose and a single oral 4 g dose administered as granules for oral suspension in healthy male and female subjects
PK parameter of zoliflodacin : Tmax | Day 3
  Tmax (the elapsed time from dosing at which Cmax was apparent) of zoliflodacin after a single oral 3 g dose and a single oral 4 g dose administered as granules for oral suspension in healthy male and female subjects
PK parameter of zoliflodacin : AUC | Day 3
  Area Under the Curve of zoliflodacin after a single oral 3 g dose and a single oral 4 g dose administered as granules for oral suspension in healthy male and female subjects
PK parameter of zoliflodacin : T1/2 | Day 3
  the apparent elimination half-life of zoliflodacin after a single oral 3 g dose and a single oral 4 g dose administered as granules for oral suspension in healthy male and female subjects

SECONDARY OUTCOMES:
safety and tolerability of zoliflodacin | end of study
  safety and tolerability of zoliflodacin after a single oral 3 g dose and a single oral 4 g dose administered as granules for oral suspension in healthy male and female subjects
relative bioavailability (Cmax) of zoliflodacin in the fed and fasted states | Day 3
  To determine the maximum observed concentration (Cmax) of zoliflodacin in the fed and fasted states
relative bioavailability (AUC) of zoliflodacin in the fed and fasted states | Day 3
  To determine the Area Under the Curve (AUC) of zoliflodacin in the fed and fasted states
zoliflodacin effect on QT intervals | Day 2
  To collect 12-lead Holter recordings to assess QTcP, QTcF, QT intervals corrected with Bazett's formula

CONTACTS AND LOCATIONS:
Overall Officials: Juan Perez-Morales, MD, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Miami, Florida, United States